CLINICAL TRIAL: NCT02396238
Title: Scleroderma Treatment With Celution Processed Adipose Derived Regenerative Cells (STAR): A Randomized, Double-Blind, Placebo-Controlled Trial With Incomplete Crossover
Brief Title: Scleroderma Treatment With Celution Processed Adipose Derived Regenerative Cells (STAR)
Acronym: STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cytori Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STAR Trial
Record Dates: First submitted 2015-03-12; First posted 2015-03-24 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-06

CONDITIONS: Scleroderma; Systemic Sclerosis; Raynaud Phenomena; Raynaud's Disease
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic; Raynaud Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adipose Derived Regenerative Cells (Experimental): Adipose Derived Regenerative Cells (ADRCs) processed by the Celution Device 40,000,000 ADRCs administered in 2 injections per digit on both hands.
  Interventions: Device: Celution Device
- Placebo (Placebo Comparator): Sterile Lactated Ringers Solution mixed with small amount of study subject's own freshly drawn blood and administered in 2 injections per digit on both hands.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Celution Device — ADRCs prepared using the investigational Celution Device
  Arms: Adipose Derived Regenerative Cells
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the safety and efficacy of the Celution Device in the processing of an autologous graft consisting of adipose derived regenerative cells (ADRCs) in the treatment of hand dysfunction due to scleroderma.

DETAILED DESCRIPTION:
The STAR Trial is a prospective, randomized, multi-center device trial intended to assess safety and efficacy of subcutaneous administration of Celution processed ADRCs into fingers of patients with hand dysfunction due to scleroderma.

Following informed consent and screening evaluations, eligible subjects will undergo pre-operative testing. Subjects will then undergo fat harvest through small volume liposuction under local anesthesia. Lipoaspirate will be processed in the Celution System to isolate and concentrate ADRCs for immediate subcutaneous administration under local anesthesia. Subjects will be randomly assigned to receive ADRCs (40 million cells) or a visually-matched placebo in a 1:1 ratio. All subjects will receive subcutaneous administration of test substance (ADRC or placebo) into all fingers of both hands. Following completion of all 48 week visits and database lock, placebo treated subjects will be offered treatment with their ADRCs cells should they continue to qualify according to the inclusion/exclusion criteria and should they wish to be treated with ADRCs and agree to the fat harvest procedure.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males or females ≥ 18 and ≤ 70 years of age
2. Diagnosis of diffuse cutaneous scleroderma (duration > 5 years) or limited cutaneous scleroderma.
3. Cochin score ≥ 20 units
4. Ability to safely undergo liposuction
5. Symptoms consistent with Raynaud's Phemomena
6. Compliant with standard preventative recommendations

Key Exclusion Criteria:

1. Body Mass Index < 18 kg/m2
2. Active infection in any finger during screening period or infection in any finger requiring antibiotics in the 30 days prior to the Screening Visit
3. Active infection at the potential site(s) of fat harvest during the screening period
4. Contractures of any finger or ulceration at point of injection precluding completion of injection procedure
5. Amputation of any finger proximal to the proximal interphalangeal joint or any amputation in more than one finger
6. Diagnosis of Rheumatoid Arthritis
7. Inflammatory arthritis of the hand, including significant osteoarthritis, that is not due to scleroderma or significant acute inflammation in the hand that is due to scleroderma, as per the investigator's clinical judgment
8. Oral cyclophosphamide exceeding 2 mg/kg/day, any intravenous cyclophosphamide, methotrexate exceeding 25 mg/week, mycophenolate mofetil exceeding 3 gm/day, hydoxychloroquine exceeding 7 mg/kg/day or azathioprine exceeding 300 mg/day or any other immunosuppressive medication in the 90 days prior to the Screening Visit

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-05-15 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2018-05-22 (Actual)

PRIMARY OUTCOMES:
Cochin score | 24 Weeks

SECONDARY OUTCOMES:
Cochin score | 48 Weeks
Raynaud's Condition Score | 24 Weeks
Scleroderma Health Assessment Questionnaire (SHAQ) | 24 Weeks

OTHER OUTCOMES:
Cochin Score | up to 48 Weeks
Raynaud's Condition Score | up to 48 Weeks
Scleroderma Health Assessment Questionnaire (SHAQ) | up to 48 Weeks
Physician and Patient Global Assessment | up to 48 Weeks
Hand Mobility in Scleroderma (HAMIS) | up to 48 Weeks
Digital ulcer count | up to 48 Weeks
Modified Rodnan Score | up to 48 Weeks
Grip strength and pinch strength | up to 48 Weeks
Finger circumference (with hand volume) | up to 48 Weeks
1st corner distance and sum of 2nd, 3rd and 4th corner distances | up to 48 Weeks
The EuroQOL five dimensions questionnaire (EQ-5D) | up to 48 Weeks
Adverse events, Serious Adverse Events | up to 48 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven Kesten, MD, Study Director — Cytori Therapeutics
Locations (19):
- United States (19):
  - Arizona Arthritis and Rheumatology Research, PLLC, Phoenix, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Arthritis Associates of Southern California, Los Angeles, California
  - UCLA David Geffen School of Medicine, Los Angeles, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - Heartland Research Associates, Wichita, Kansas
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - West Michigan Rheumatology, PLLC, Grand Rapids, Michigan
  - Center For Pharmaceutical Research, Kansas City, Missouri
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Hospital for Special Surgery, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Houston Medical School, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khanna D, Caldron P, Martin RW, Kafaja S, Spiera R, Shahouri S, Shah A, Hsu V, Ervin J, Simms R, Domsic RT, Steen V, Hummers LK, Derk C, Mayes M, Chatterjee S, Varga J, Kesten S, Fraser JK, Furst DE. Adipose-Derived Regenerative Cell Transplantation for the Treatment of Hand Dysfunction in Systemic Sclerosis: A Randomized Clinical Trial. Arthritis Rheumatol. 2022 Aug;74(8):1399-1408. doi: 10.1002/art.42133. Epub 2022 Jun 27. PMID 35358372